CLINICAL TRIAL: NCT03895619
Title: Getting to Zero: Safer Conception Programming to Eliminate Sexual and Perinatal HIV Transmission Among HIV Sero-different Couples in Uganda
Brief Title: Getting to Zero: Safer Conception Programming Among HIV Sero-different Couples in Uganda
Acronym: G2Z
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Mbarara University of Science and Technology (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angela Kaida, Associate Professor, Simon Fraser University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018s0272
Record Dates: First submitted 2018-10-29; First posted 2019-03-29 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Proof of Concept Research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men living with HIV (Experimental): Uptake of safer conception strategies among men living with HIV and/or their female partners
  Interventions: Other: Safer conception strategies

INTERVENTIONS:
Other: Safer conception strategies — Individuals and couples adopt safer conception strategies including HIV-serostatus disclosure to partner, ART uptake and adherence and HIV-RNA suppression, STI testing and treatment, timing condomless sex to peak fertility, partner ARV use (ART if living with HIV, PrEP if HIV negative), and contraception until ready to conceive.

SUMMARY:
Despite effective strategies to reduce periconception HIV transmission, there are few services to support people living with or affected by HIV to use these methods. In particular, there is a lack of safer conception services focused on engaging men living with HIV. Given known gender inequities in childbearing decision-making and HIV risk, it is critical that safer conception services deliver programming that engages men living with HIV and their HIV sero-different partners. The Healthy Families program, based at the ISS Clinic at Mbarara Regional Referral Hospital, offers client-centered safer conception care to help HIV-affected individuals and couples meet reproductive goals. This care supports clients to leverage personal motivations and partner and social supports to overcome structural barriers and use Antiretroviral Therapy (ART), adopt other HIV-prevention strategies, and remain in care. This pilot study (the 'Getting to Zero' study) will assess uptake and experiences of safer conception care among 50 men living with HIV and their HIV sero-different partners. Investigators will also assess men's retention in HIV care and HIV transmission risk to partners and infants. This is a one-year mixed-methods prospective pilot research study, which will use electronic chart review data, longitudinal survey data (from the male index and female partner participant), and qualitative data from in-depth semi-structured interviews to meet study objectives. By demonstrating safer conception uptake and impact on HIV transmission risks to partners and infants, investigators aim to inform HIV and reproductive health policy in Uganda and globally.

DETAILED DESCRIPTION:
The Healthy Families safer conception program, based at the ISS Clinic at Mbarara Regional Referral Hospital (MRRH), offers client-centered care to help HIV-affected individuals and couples meet reproductive goals. This care supports clients to leverage personal motivations and partner and social supports to overcome structural barriers and use ART, adopt other HIV-prevention strategies, and remain in care. This pilot study (the 'Getting to Zero' study) will assess uptake and experiences of safer conception care among men living with HIV and their HIV sero-different partners, and will assess retention in care and HIV transmission risk to partners and infants.

There are six linked objectives in this study:

1. To assess uptake of safer conception strategies among men living with HIV and/or their female partners overall, and by specific HIV prevention strategies.

   Hypothesis 1: Investigators hypothesize that offering comprehensive safer conception services within HIV care will increase uptake of HIV prevention strategies among both male and female HIV-affected participants (including ART initiation, adherence, and HIV-RNA viral suppression in the partner living with HIV, HIV-serostatus disclosure, knowledge of partner's HIV-serostatus, Sexually Transmitted Infections (STI) testing and treatment, sexual behaviour (i.e., delaying condomless sex until HIV-infected partner is virally suppressed), and partner HIV testing and ARV use (PrEP or ART).
2. Among men living with HIV and their partners, to assess socio-demographic, relationship, structural, and clinical factors associated with uptake of safer conception strategies.

   Hypothesis 2: Investigators hypothesize that uptake will be associated with more equitable relationship power and dynamics, lower HIV-related stigma, higher social support, and other socio-structural determinants of health.
3. To assess retention in HIV care among men living with HIV engaged in the safer conception intervention.

   Hypothesis 3: Investigators hypothesize that men living with HIV who are engaged in the safer conception intervention will be better retained in HIV care over nine months relative to men receiving care at the ISS clinic, but who are not enrolled in the safer conception program.
4. To assess periconception HIV transmission incidence among HIV-affected individuals and couples where the male partner is living with HIV and engaged in the safer conception intervention;

   Hypothesis 4: Among HIV-affected individuals and couples successfully engaged in the safer conception intervention, investigators hypothesize no (within-couple) cases of periconception-related HIV transmission.
5. To assess pregnancy and HIV incidence and outcomes among female partners of men living with HIV engaged in the intervention.

   Hypothesis 5: Of pregnancies ending in live birth, investigators hypothesize <2% incidence of perinatal HIV transmission among infants born to couples successfully engaged in the intervention.
6. To explore the acceptability and barriers/facilitators of the safer conception intervention among a sub-set of men living with HIV and their HIV sero-different partners.

Hypothesis 6: This is qualitative objective without pre-specified hypotheses.

This study will be conducted at the ISS Clinic in the Mbarara Regional Referral Hospital (MRRH) in Mbarara, Uganda.

This mixed-methods prospective pilot research study includes electronic chart review data, longitudinal survey data (from the male index and female partner participant), and qualitative data from in-depth semi-structured interviews. All of the study efforts will be conducted via the Immune Suppression Syndrome (ISS) Clinic in the Mbarara Regional Referral Hospital in Mbarara, Uganda. The ISS clinic is an IeDEA networks site with a high-quality clinical database. In December 2016, the ISS clinic initiated a safer conception program called the Healthy Families program, which provides counselling and clinical care for HIV-affected individuals and couples who desire pregnancy.

The target population for the Getting to Zero study is men living with HIV with HIV sero-different partners (defined as partners who are HIV-negative or HIV status unknown), who report personal and/or partner pregnancy desire in the next year. Participants will be recruited via information sessions held at the Healthy Families program as well as at the ISS Clinic, MRRH HIV counselling and testing sites, referrals from regional healthcare providers, and via community outreach efforts.

This pilot study aimed at demonstrating proof-of-concept aims to enroll 50 index participants and all female partners. Investigators anticipate, however, enrolling 25 female partners.

The target population for the Getting to Zero study is men living with HIV with HIV sero-different partners (defined as partners who are HIV-negative or HIV status unknown), who report personal and/or partner pregnancy desire in the next year. Participants will be recruited via information sessions held at the Healthy Families program as well as at the ISS Clinic, MRRH HIV counselling and testing sites, referrals from regional healthcare providers, and via community outreach efforts. After providing informed consent, participants will be asked to complete an interviewer-administered questionnaire detailing use of HIV prevention strategies as well as socio-demographic information, partnership dynamics, pregnancy intentions and desires, sexual and reproductive behaviours and history, HIV medical history, mental health, experiences of violence, HIV-related stigma, and social support.

Following the questionnaire, the participant (and his partner if she is present) will be offered safer conception services at the Healthy Families clinic, which includes an up to 30-minute counseling session. Counseling sessions incorporate education and some problem-solving support to help individuals and couples adopt safer conception strategies including HIV-serostatus disclosure to partner, ART uptake and adherence and HIV-RNA suppression, STI testing and treatment, timing condomless sex to peak fertility, partner ARV use (ART if living with HIV, PrEP if HIV negative), and contraception until ready to conceive. In addition, (1) all female partners are offered beta hcg pregnancy testing; (2) all HIV-negative participants are offered HIV counselling and testing; (3) all participants will complete testing for STIs (Neisseria gonorrhoeae, Chlamydia trachomatis, and Trichomonas vaginalis) via GeneXpert. Index participants will also complete testing for syphilis using Bioline testing (treponeme specific) followed by RPR confirmatory testing (non-treponeme specific); and (4) all participants living with HIV will also complete laboratory testing to assess HIV-RNA suppression.

Participants will be offered the safer conception counselling and clinical services at enrollment, 3-months (3M), and 6-months (6M), with two exceptions. First, STI testing will only be offered at the baseline visit for male participants only and subsequent follow-up visits will employ syndromic STI management, which is standard of care at the Healthy Families program. Second, participants will complete HIV-RNA suppression testing at enrolment and 6M.

Male participants will be asked for their consent for the study team to contact their female partners to assess eligibility, interest, and willingness to participate in the study. If he consents for the study team to contact his partner, he will be given an information letter to give to her describing the study purpose and procedures. Once consented, partners will be invited to safe conception counselling sessions as well as to participate in an individual in-depth interview to explore acceptability and barriers/facilitators of the Healthy Families program.

At enrollment and all Healthy Families program follow-up visits (3M and 6M):

1. all female partners will be offered pregnancy testing via urine beta hcg testing. Results will be available within 3-5 minutes of testing. Women who test positive for pregnancy will be referred to appropriate antenatal care.
2. all participants who are not known to be HIV-positive will be offered HIV counselling and testing. Individuals confirmed HIV-positive will receive post-test counselling and be referred for appropriate HIV care.
3. all male participants will undergo objective STI testing at enrollment with same-day pathogen-specific treatment provided for the tested individual as well as to partners. Testing for Neisseria gonorrhoeae, Chlamydia trachomatis, and Trichomonas vaginalis will be done via GeneXpert. Participants will also complete testing for syphilis using Bioline testing (treponeme specific) followed by RPR confirmatory testing (non-treponeme specific). Symptomatic male patients will be treated as per national STI syndromic management guidelines. Male participants will be given the same course of treatment to take home to their female partners.
4. all participants living with HIV will also complete laboratory testing to assess HIV-RNA suppression at baseline and 6M.

The procedures described are consistent with usual clinical management of HIV-affected individuals/couples receiving care at the Healthy Families Clinic (i.e., are part of usual clinical management).

ELIGIBILITY:
Inclusion Criteria:

For enrollment in the Getting to Zero study, eligibility criteria for the index participant include the following:

1. Identify as male
2. HIV-positive
3. Report personal or partner desire to have a child in the next year
4. Identified pregnancy partner is reported to be HIV-negative or he doesn't know her HIV serostatus.
5. Aged 18 years or older.
6. Be naïve to the Healthy Families program.
7. Live within 60km of the ISS clinic and not planning to relocate to an area incompatible with an ability to attend the clinic over a 1 year follow-up period.
8. Able and willing to participate in the informed consent process.

Men living with HIV enrolled in the Getting to Zero study (index participants) will be asked for their consent to contact their partners to determine eligibility, interest, and willingness to participate in the Getting to Zero study. Partner participants must meet the following inclusion criteria:

1. Identify as a partner of an enrolled male Getting to Zero participant
2. Aged 18 years or older
3. Able and willing to participate in the informed consent process.

These participants will be referred to as the "partner". If the female partner is identified as HIV-positive after the male index participant enrolls in the Getting to Zero study, both partners remain eligible to participate.

Exclusion Criteria for Index Participant:

1. Identify as female
2. HIV-negative
3. Does not report personal or partner desire to have a child in the next year
4. Identified pregnancy partner is reported to be HIV-positive
5. Under age 18 years.
6. Be a patient of the Healthy Families program.
7. Live greater than 60km of the ISS clinic and planning to relocate to an area incompatible with attending the clinic over a 1 year follow-up period.
8. Unable and unwilling to participate in the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of HIV infected men and their female partners attending Safer Conception Counselling Sessions and choosing a safer conception strategy that meets their needs | 1.5 year
  We will document the number of participants who return to their clinic with their female pregnancy partner to attend Safer Conception Counselling. We will also document the type of strategy chosen.

SECONDARY OUTCOMES:
Types of factors contributing to uptake of safer conception strategies among men living with HIV | 1.5 year
  The reasons why men chose to use safer conception strategies will be better understood using unadjusted and adjusted logistic regression models (with 95% confidence intervals)
Number of men living with HIV retained in care who are part of the safer conception intervention. | 1.5 year
  Will use Kaplan-Meier methods to measure time to index loss from care
HIV transmission incidence among HIV-affected individuals and couples where the male partner is living with HIV and engaged in the safer conception intervention. | 1.5 year
  Will use Kaplan-Meier methods to measure partner HIV-seroconversion.
Periconception HIV transmission incidence among HIV-affected individuals and couples. | 1.5 year
  Cumulative incidence of pregnancy will be calculated as the total number of pregnancies over the follow-up period by person-years of follow-up.
HIV incidence among female partners of men living with HIV engaged in the safer conception intervention. | 1.5 year
  Will analyze interview data using content analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Immune Suppression Syndrome (ISS) Clinic at the Mbarara Regional Referral Hospital (MRRH), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided